CLINICAL TRIAL: NCT00751283
Title: Minnow Medical GRST Peripheral Catheter System First-in-Man Study Radiofrequency for the Treatment of Peripheral Vascular Occlusive Disease of the Lower Extremities
Brief Title: Radiofrequency for the Treatment of Peripheral Vascular Occlusive Disease of the Lower Extremities
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Data was inconclusive
Sponsor: Vessix Vascular, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DR0052
Record Dates: First submitted 2008-09-09; First posted 2008-09-11 (Estimated); Last update posted 2013-08-14 (Estimated); Status verified 2013-08

CONDITIONS: Peripheral Vascular Disease
MeSH Terms: conditions — Peripheral Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): GRST Peripheral Catheter System
  Interventions: Device: GRST Peripheral Catheter System

INTERVENTIONS:
Device: GRST Peripheral Catheter System — Treatment to dilate stenoses and reduce plaque in treated vessels

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of the Minnow Medical GRST Peripheral Catheter System in the treatment of new lesions in the superficial femoral artery or the popliteal artery.

ELIGIBILITY:
Inclusion Criteria:

* Patient is ≥18 years of age
* Patient is Rutherford category 2-4
* De novo lesion in the SFA or popliteal artery with a diameter stenosis ≥50%
* Target lesion is a de novo occlusion that can be successfully pre-dilated resulting in a lesion of <99%
* Target lesion stenosis has a length of ≤100 mm based on visual assessment
* Target vessel reference diameter is ≥3.0 mm and ≤7.0 mm based on visual assessment
* Angiographic evidence of distal runoff defined as minimum one (1) patent tibial artery with a straight flow to the foot
* Patient is willing and able to provide written informed consent prior to any study specific procedure
* Patient is willing and able to comply with specified follow-up evaluations at the specified times

Exclusion Criteria:

* Any prior intervention in the intended target lesion including 10 mm proximal or distal from the intended treatment area
* Evidence of thrombus in the target vessel
* Prior ipsilateral or contralateral lower limb arterial bypass
* Treatment of ipsilateral lesions during the index procedure or planned treatment after the index procedure
* Target lesion is severely calcified
* Any known allergies and / or intolerances to the following: ASA, Clopidogrel, Heparin, contrast agents (that cannot be adequately pre-medicated).
* Any planned surgery within 30 days of the study procedure.
* Renal failure (serum creatinine > 2.0 mg/dL)
* Female with childbearing potential without a negative pregnancy test
* Patient has had an organ transplant
* Patient is currently participating in an investigational drug or device study which has not reached the primary endpoint yet or which clinically interferes with the endpoints of this study
* In the investigator's opinion, the patient has a severe co-morbid condition(s) that could limit the ability to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-08; Primary Completion 2010-11 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Major adverse clinical events rate | Up to 30 days

SECONDARY OUTCOMES:
Binary restenosis | 30 days, 3 months, 6 months
Target lesion revascularization | 30 days, 3 months, 6 months
Amputation rate | 30 days, 3 months, 6 months
Technical success | Treatment
Serious adverse events rate, including major adverse clinical events | 30 days, 3 months, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Dierk Scheinert, MD, Principal Investigator — Universität Leipzig Herzzentrum